CLINICAL TRIAL: NCT00452647
Title: Comparison of Blood Pressure Throughout Pregnancy
Status: Terminated | Type: Observational
Why Stopped: data did not indicate any meaningful information
Sponsor: Drexel University College of Medicine (Other)
Responsible Party: Principal Investigator, Marcus Zebrower, Investigator, Drexel University
Organization: Drexel University (Other)
Other Study IDs: 16807
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Condition: No specific disease is being studied, few procedures are excluded.; Focus: To obtain blood pressure data and detect any trends to a statistically significant degree.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to observe and analyze variation of diastolic blood pressure measurements at third trimester of pregnancy and when they present for delivery in comparison to healthy volunteers.

When patients present for delivery, we expect blood pressure to be lower than normal. However this is not the case. We aim to determine where this trend occurs throughout to duration of pregnancy, and propose possible explanation as to the source of this event.

After discharge, the information recorded includes each patient's blood pressure upon admission to the labor floor, and several blood pressure measurements from prior clinical visits.

ELIGIBILITY:
Inclusion Criteria:

* Females age 18-40
* Parturients who present for delivery who are not yet in labor

Exclusion Criteria:

* Patients with hypertension, cardiac disease, diabetes, or thyroid disorders
* Parturients who are already in labor upon presentation to the labor floor

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Population defined as parturients who present for delivery. See Eligibility Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Measurment of blood pressure throught pregnancy | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jay Horrow, MD, Study Chair — Drexel University College of Medicine
Locations (1):
- Hahnemann University Hospital, Philadelphia, Pennsylvania, United States